CLINICAL TRIAL: NCT02776592
Title: Nutritive Effects of a Cow's Milk Based Formula Fed to Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: Federal University of Bahia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 6036
Record Dates: First submitted 2016-05-12; First posted 2016-05-18 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Child Nutrition Sciences
Keywords: Healthy Children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): A cow's milk-based formula with added nutrients
  Interventions: Other: Cow's milk-based formula with added nutrients
- Control (Active Comparator): A cow's milk-based formula
  Interventions: Other: Cow's milk-based formula

INTERVENTIONS:
Other: Cow's milk-based formula with added nutrients
  Arms: Experimental
Other: Cow's milk-based formula
  Arms: Control

SUMMARY:
This study aims to determine if a cow's milk-based formula with added nutrients has an effect on memory, reaction time, strategy or other cognitive development indicators in children 4-5 years of age.

DETAILED DESCRIPTION:
This study aims to determine if a cow's milk-based formula with added nutrients has an effect on memory, reaction time, strategy or other cognitive development indicators in children 4-5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Health child, 4-5 years of age
* Born as full-term (Gestational age of 37-42 weeks)
* Consumed cow's milk or a cow's milk-based beverage during the 48 hours prior to the baseline visit
* Parents or legal guardian agrees not to feed child any food products or supplements containing probiotics or prebiotics
* Signed informed consent

Exclusion Criteria:

* History or known or suspected cow milk protein intolerance
* Child who has received any food product ot supplement containing probiotics or prebiotics (with the exception of yogurt) in the 15 days prior to the baseline visit
* Serious concurrent illness that will interfere in the general management of the child
* History of underlying metabolic or chronic disease, congenital malformation, or immunocompromised
* Child's z-score of weight for height at baseline is < -3 according to WHO criteria

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 199 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2016-12-23 (Actual); Study Completion 2016-12-23 (Actual)

PRIMARY OUTCOMES:
Change in Working Memory Capacity | Up to 24 weeks
  Recall of variable sequences

SECONDARY OUTCOMES:
Change in Motor Response Speeds | Up to 24 weeks
Change in Mental Response Speeds | Up to 24 weeks
Change in Retention of Visual Information | Up to 24 weeks
Change in Manipulation of Visual Information | Up to 24 weeks
Change in Child Behavior Checklist | Up to 24 weeks
  Assessment of adaptive function
Stool Consistency Assessment | 24 weeks
Systemic antibiotic Usage | 24 weeks
Missed days due to illness | 24 weeks
Body Weight | 24 weeks
Height | 24 weeks
Study Product Intake Assessment | 24 weeks
Complete Blood Count (CBC) | Up to 24 weeks
Blood Fatty Acids | Up to 24 weeks
Metabolite Biomarkers | Up to 24 weeks
Serum Phospholipids | Up to 24 weeks
Immune Markers | Up to 24 weeks
Medically-confirmed adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jon Vanderhoof, M.D., Study Director — Mead Johnson Nutrition
Locations (1):
- Research Center Fima Lifshitz - Federal University of Bahia, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No